CLINICAL TRIAL: NCT00796679
Title: A Prospective, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy of Oral Paricalcitol in Retarding Cardiac Hypertrophy, Reducing Inflammation and Atherosclerosis in Stage 3 - 5 Chronic Kidney Disease
Brief Title: Oral Paricalcitol in Stage 3 - 5 Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Dr., The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A10-003
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease
Keywords: paricalcitol; chronic kidney disease; cardiac hypertrophy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiomegaly | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): paricalcitol
  Interventions: Drug: paricalcitol
- 2 (Placebo Comparator): placebo
  Interventions: Drug: paricalcitol

INTERVENTIONS:
Drug: paricalcitol — oral paricalcitol capsule 1 microgram once daily if iPTH <500pg/mL or 2 microgram once daily if iPTH >=500pg/mL. Thereafter, dose titration in 1 microgram decrement will be done based on safety reasons (that is, for low PTH or high calcium and phosphorus level). The duration of treatment will be for 1 year.
  Other Names: Zemplar

SUMMARY:
The purpose of this study is to test the hypothesis that selective vitamin D receptor activation reduces left ventricular hypertrophy and ameliorates inflammation and atherosclerosis in stage 3 -5 chronic kidney disease.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality and morbidity in patients with chronic kidney disease. According to a previous study, only 15.6% of the patients beginning dialysis therapy had a normal echocardiogram, with left ventricular hypertrophy, left ventricular dilatation and systolic dysfunction occurring in 40.7%, 28% and 15.6% of patients, respectively. In addition, these patients are at an accelerated risk of developing atherosclerosis. The Kidney Disease Outcome Quality Initiative guideline recently raised concerns of a high prevalence of vitamin D deficiency in chronic kidney disease patients not yet requiring dialysis treatment. In addition, very recent data suggested that vitamin D deficiency is an important predictor of mortality in end-stage renal disease patients. Furthermore, hemodialysis patients treated with paricalcitol, a selective vitamin D receptor activator, showed a significantly lower risk of cardiovascular death than those not receiving vitamin D therapy. A number of studies also showed positive benefit of vitamin D receptor activator treatment on regression of left ventricular hypertrophy in dialysis patients. However, there is so far no data in patients with stage 3 and 4 chronic kidney disease where a high prevalence of vitamin D deficiency and cardiac hypertrophy has been reported.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage 3 -5 chronic kidney disease (that is, eGFR < 60 ml/min per 1.73m2) diagnosed for more than 2 months and not expected to start dialysis within the next 12 months, and
* Patient with screening echocardiography showing evidence of left ventricular hypertrophy
* Patient has not received vitamin D therapy in the previous 4 weeks
* For entry into the Treatment Phase, the subject must have:

  * screening iPTH >= 55 pg/ml or 5.8pmol/L (determined by the Nichols second-generation assay or similar assay)
  * serum calcium < 10.2 mg/dL (2.55 mmol/L)
  * serum phosphorus =< 5.2mg/dL (1.68mmol/L)
  * Ca*P product < 54 mg2/dL2 (4.36mmol2/L2)
  * If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or is of childbearing potential and practicing birth control measures.
* Patients who provide informed consent for the study

Exclusion Criteria:

* Patient with a history of an allergic reaction or significant sensitivity to vitamin D or vitamin D related compounds.
* Patient with history of renal stones
* Patient with current malignancy
* Patients with clinically significant gastrointestinal disease or liver disease
* Patient with acute renal failure in the recent three months
* Patient with a history of drug or alcohol abuse within six months prior to the screening phase
* Patient is known to be human immunodeficiency virus (HIV) positive.
* Patient with evidence of poor compliance with diet and medication.
* Patient currently receiving medications that may affect calcium, phosphorus metabolism such as calcitonin, cinacalcet, bisphophonates or vitamin D compounds (other than study drug), or other drugs that may affect calcium or bone metabolism, other than females on stable estrogen and/or progestin therapy.
* Patients with active granulomatous disease
* Patient with pregnancy
* Patients currently receiving glucocorticoid steroid or other immunosuppressive treatment or had been administered glucocorticoid or other immunosuppressive treatment for more than 14 days within recent 6 months.
* Patients with contraindication for MRI examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass index determined by MRI | 1 year

SECONDARY OUTCOMES:
Change in left atrial and ventricular volumes, systolic and diastolic function, carotid intima-media thickness, flow mediated dilation, pulse wave velocity, serum inflammatory and cardiac biomarkers, intact PTH, 24-hour urine protein and renal function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD, FRCP, Principal Investigator — Queen Mary Hospital, University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - University of Hong Kong, Queen Mary Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang AY, Fang F, Chan J, Wen YY, Qing S, Chan IH, Lo G, Lai KN, Lo WK, Lam CW, Yu CM. Effect of paricalcitol on left ventricular mass and function in CKD--the OPERA trial. J Am Soc Nephrol. 2014 Jan;25(1):175-86. doi: 10.1681/ASN.2013010103. Epub 2013 Sep 19. PMID 24052631